CLINICAL TRIAL: NCT05606939
Title: The Role of Intestinal Ultrasound in Monitoring the Response to Biological Therapy in Patients With Ulcerative Colitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Abanoub Ayoub Melk, resident doctor at tropical medicine and gastroenterology, Assiut University
Other Study IDs: IUS in ulcerative colitis
Record Dates: First submitted 2022-08-03; First posted 2022-11-07 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: intestinal ultrasound — All patients will be evaluated using intestinal ultrasound with special emphasis on intestinal wall thickness as well as stratification and Visualization of the vascularization of the bowel using color Doppler sonography also visualization of motility.
  Findings of intestinal ultrasound will be compared regrading colonoscopic findings

SUMMARY:
In this study, the investigators aim to evaluate the role of intestinal ultrasound in evaluation of the therapeutic response to biological therapy in patient with ulcerative colitis

DETAILED DESCRIPTION:
Ultrasound examination is an easily accessible, non-invasive, radiation-free technique, and cheap imaging modality that is often chosen as the first diagnostic method in gastroenterology disease.

performance of bowel ultrasound use of two different probes: low-frequency convex probe (3.0-3.5 MHz) and high-frequency linear probe (5-17 MHz) .

Inflammatory bowel disease (IBD) is a chronic inflammatory disease of the gastrointestinal tract, which clinically contains Crohn's disease, ulcerative colitis, and other conditions. IBD is characterized by episodes of abdominal pain, diarrhea, bloody stools, weight loss, and the influx of neutrophils and macrophages that produce cytokines, proteolytic enzymes

Intestinal ultrasound has been shown to have high sensitivity and specificity in the detection or exclusion of intestinal inflammatory activity in IBD. advantages of intestinal ultrasound over other imaging modalities include non-invasiveness, rapid availability and low costs ,evaluation of bowel wall thickness, as well as stratification that reflects alterations in histopathology ulcerative colitis (UC). Visualization of the vascularization of the bowel using color Doppler sonography and, direct visualization of motility.

A study done : IUS is preferred for monitoring the disease course and for assessing short-term treatment response. Found that monitoring bowel wall thickening (BWT) alone has the potential to predict the therapeutic response.The primary therapeutic goal in UC is to induce and maintain long-term disease remission; however, there is no single treatment pathwayguidelines recommend the use of either conventional therapies (i.e., aminosalicylates ..etc)Or the use of biologic therapies ( infliximab.)

ELIGIBILITY:
Inclusion Criteria:

* Any patient above age of 18 years old and diagnosed to have UC and whom not responding to conventional medical therapy and eligible for biological therapy will be recruited in this study

  * moderate to severe UC patients
  * immunosuppressant or corticosteroid refractory disease
  * those with intolerance or contraindication to conventional therapies are eligible to be treated with biological therapy

Exclusion Criteria:

* Patients with UC who are under age of 18 years' old
* Patients with UC who aren't eligible to biological therapy
* patients with complication of UC(fistula , intestinal obstruction , intestinal perforation ,……)
* Patient refuse to participate in the study.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any patient above age of 18 years old and diagnosed to have UC and whom not responding to conventional medical therapy and eligible for biological therapy will be recruited in this study
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-03-12 (Estimated)

PRIMARY OUTCOMES:
the role of intestinal ultrasound in evaluation of the therapeutic response to biological therapy in patient with ulcerative colitis | Baseline , 2 weeks , 6 weeks
  All patients will be evaluated using intestinal ultrasound with special emphasis on intestinal wall thickness in mm as well as stratification normal or dirupted and Visualization of the vascularization (normal decrease or increased) of the bowel using color Doppler sonography also visualization of motility (normal , increased or decreaed) Findings of intestinal ultrasound will be compared regrading colonoscopic findings to evaluate the response to biological therapy through IUS

REFERENCES:
- [Background] Zakeri N, Pollok RC. Diagnostic imaging and radiation exposure in inflammatory bowel disease. World J Gastroenterol. 2016 Feb 21;22(7):2165-78. doi: 10.3748/wjg.v22.i7.2165. PMID 26900282
- [Background] Atkinson NSS, Bryant RV, Dong Y, Maaser C, Kucharzik T, Maconi G, Asthana AK, Blaivas M, Goudie A, Gilja OH, Nuernberg D, Schreiber-Dietrich D, Dietrich CF. How to perform gastrointestinal ultrasound: Anatomy and normal findings. World J Gastroenterol. 2017 Oct 14;23(38):6931-6941. doi: 10.3748/wjg.v23.i38.6931. PMID 29097866
- [Background] Jauregui-Amezaga A, Rimola J. Role of Intestinal Ultrasound in the Management of Patients with Inflammatory Bowel Disease. Life (Basel). 2021 Jun 23;11(7):603. doi: 10.3390/life11070603. PMID 34201630
- [Background] Novak KL, Nylund K, Maaser C, Petersen F, Kucharzik T, Lu C, Allocca M, Maconi G, de Voogd F, Christensen B, Vaughan R, Palmela C, Carter D, Wilkens R. Expert Consensus on Optimal Acquisition and Development of the International Bowel Ultrasound Segmental Activity Score [IBUS-SAS]: A Reliability and Inter-rater Variability Study on Intestinal Ultrasonography in Crohn's Disease. J Crohns Colitis. 2021 Apr 6;15(4):609-616. doi: 10.1093/ecco-jcc/jjaa216. PMID 33098642